CLINICAL TRIAL: NCT02618148
Title: The Natural Ingredients and Artificial Made Ready, a Good Combination Reduced the Risk of Thrombosis, Concerns With Their Use of HRT
Brief Title: Hormone Estradiol Replacement Therapy Additional Herbals
Acronym: WH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Trieu, Nguyen Thi, M.D. (Individual)
Responsible Party: Principal Investigator, Nguyen Thi Trieu, MD, Sponsor, Trieu, Nguyen Thi, M.D.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Estrogen Herbals
Record Dates: First submitted 2015-11-14; First posted 2015-12-01 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Menopause

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESTROGEN HERBALS 21 (Experimental): Used for women who wish to monthly menstruation
  Applies to the following strengths:
  17β-estradiol 1.5mg/24 hours x 21 days, stop drinking for 7 days. Progesterone 5mg/24 hours x 10 days, stop drinking for 7 days. Garlic oil 30mg/24 hours x 28 days. Enzyme nattokinase 300 FU x 24 hours x 28 days.
  Interventions: Drug: ESTROGEN HERBALS 21
- ESTROGEN HERBALS 28 (Experimental): Used for women who do not wish to monthly menstruation
  Applies to the following strengths:
  17β-estradiol 1.5mg/24 hours x 28 days. Garlic oil 30mg/24 hours x 28 days. Enzyme nattokinase 300 FU x 24 hours x 28 days.
  Interventions: Drug: ESTROGEN HERBALS 28

INTERVENTIONS:
Drug: ESTROGEN HERBALS 21 — Applies to the following strengths:
  17β-estradiol 1.5mg/24 hours x 21 days, stop drinking for 7 days. Progesterone 5 mg/24 hours x 10 days, stop drinking for 7 days. Garlic oil 30mg/24 hours x 28 days. Enzyme nattokinase 300 FU x 24 hours x 28 days.
  Other Names: EPGANA 21
  Arms: ESTROGEN HERBALS 21
Drug: ESTROGEN HERBALS 28 — Applies to the following strengths:
  17β-estradiol 1.5mg/24 hours x 28 days. Garlic oil 30mg/24 hours x 28 days. Enzyme nattokinase 300 FU x 24 hours x 28 days.
  Other Names: EPGANA 28
  Arms: ESTROGEN HERBALS 28

SUMMARY:
The purpose of this study is to determine whether Hormone Replacement Therapy (HRT), safety studies are combined with herbal (garlic oil, rutin, and nattokinase) to reduce estrogen side effects. Making it safer when an endocrine supplement is needed for estrogen deficiency symptoms in menopausal and postmenopausal women.

DETAILED DESCRIPTION:
Recent studies have proved :

-Garlic oil as garlic may reduce platelet aggregation, patients taking anticoagulant medication are cautioned about consuming garlic.

A 2013 meta-analysis concluded that garlic preparations may effectively lower total cholesterol by 11-23 mg/dL and LDL cholesterol by 3-15 mg/dL in adults with high cholesterol if taken for longer than two months. The same analysis found that garlic had a marginally positive effect on HDL cholesterol, no significant effect on blood triglyceride levels, and that garlic preparations were generally well tolerated with very few side effects.

* Nattokinase Nattō is made from fermented soybeans and has been eaten in Japan for about a thousand years. Nattō is produced by fermentation by adding the bacterium Bacillus natto to boiled soybeans. Nattokinase is produced by the bacterium acting on the soybeans . While other soy foods contain enzymes, it is only the nattō preparation that contains the specific nattokinase enzyme.
* Estradiol valerate is one of the most widely used esters of estradiol.
* Progesterone: Hormone replacement therapy. Progesterone is combined with 17-beta estradiol in the estrogen patch.

ELIGIBILITY:
Inclusion Criteria:

* Hormone replacement therapy (HRT) for oestrogen deficiency symptoms in perimenopausal and postmenopausal women.
* Prevention of osteoporosis in postmenopausal women at high risk of future fractures who are intolerant of, or contraindicated for, other medicinal products approved for the prevention of osteoporosis.

Exclusion Criteria:

* Known, past or suspected breast cancer;
* Known or suspected oestrogen-dependent malignant tumours (eg endometrial cancer);
* Undiagnosed genital bleeding;
* Untreated endometrial hyperplasia;
* Previous or current venous thromboembolism (deep venous thrombosis,pulmonary embolism)
* Known thrombophilic disorders (eg protein C, protein S, or antithrombin deficiency, see section.
* Active or recent arterial thromboembolic disease (eg angina, myocardial infarction);
* Acute liver disease, or a history of liver disease as long as liver function tests have failed to return to normal;
* Known hypersensitivity to the active substances or to any of the excipients;

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Time to Estradiol > 35 pg / ml | 1 years
  * Patients fulfilling inclusion and exclusion criteria.
  * Measure the time to Estradiol > 35 pg / ml
    * Will be divided into two groups Group (A): Females premenopausal Group (B): Females postmenopausal
    * Females premenopausal: (Reference Range: (35-525 pg/mL)
    * Females postmenopausal: (Reference Range:(0-35 pg/mL)

SECONDARY OUTCOMES:
Time to Estradiol > 35 pg / ml | 2 years
  - Measure the time to Estradiol > 70 pg /ml.

CONTACTS AND LOCATIONS:
Overall Officials: Tran Minh Cam Tu, Dr., Study Director — Nguyen Thi Trieu, Dr.
Locations (2):
- Saigon Biopharma LLC, Wilmington, Delaware, United States
- Saigon Biopharma Company Limited, Ho Chi Minh City, Vietnam

REFERENCES:
- See also: Garlic Oil — https://en.wikipedia.org/wiki/Garlic
- See also: Nattokinase — https://en.wikipedia.org/wiki/Nattokinase
- See also: Progesterone — http://www.nativeremedies.com/ailment/low-progesterone-levels-information.html
- See also: Estradiol — https://www.nhs.uk/conditions/hormone-replacement-therapy-hrt/types/